CLINICAL TRIAL: NCT01180647
Title: Extended-Release Naltrexone for Opioid Relapse Prevention Following Release From Jail
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Alkermes, Inc. (Industry); New York City Department of Health and Mental Hygiene (Other Government)
Responsible Party: Principal Investigator, Joshua D. Lee, Assistant Professor, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NYU IRB Number: 09-0372
Record Dates: First submitted 2010-08-10; First posted 2010-08-12 (Estimated); Results first posted 2016-04-07 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-03

CONDITIONS: Opiate Dependence
Keywords: Extended-release naltrexone; Prisoners; Opioid addiction prevention; Medication Treatment Alternatives; Prevention of Relapse to Opioid Addiction
MeSH Terms: conditions — Opioid-Related Disorders | interventions — vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extended-release naltrexone (XR-NTX) (Active Comparator): A single 380mg IM depot injection of XR-NTX in the week prior to release from jail. A second 380mg IM injection is offered to persons in the XR-NTX arm post-release and 4 weeks after the initial injection.
  Interventions: Drug: Extended-Release Naltrexone
- Motivational Enhancement Counseling Only (Placebo Comparator): The randomized control arm receives no medication treatment and is offered brief, two-session Motivational Enhancement counseling prior to release from jail.
  Interventions: Behavioral: Motivational Enhancement Counseling

INTERVENTIONS:
Drug: Extended-Release Naltrexone — 380mg IM XR-NTX injection one week prior to release from jail; a second XR-NTX 380mg IM injection is offered 4 weeks later (monthly).
  Other Names: Vivitrol
  Arms: Extended-release naltrexone (XR-NTX)
Behavioral: Motivational Enhancement Counseling — The randomized control arm receives no medication treatment and is offered brief, two-session Motivational Enhancement counseling prior to release from jail.
  Arms: Motivational Enhancement Counseling Only

SUMMARY:
This pilot study's primary aim is to compare rates of sustained opioid relapse, defined as self-reported opioid use >50% (>15 of 30) of days during the first 30 days following release from jail, among persons treated with XR-NTX pre-release vs. controls not receiving XR-NTX.

DETAILED DESCRIPTION:
This protocol randomizes persons soon-to-be-released from a large urban jail to treatment with extended-release naltrexone (XR-NTX), a full opioid antagonist that prevents the activity of heroin and other opioids. Investigators at NYUSOM and NYC DOHMH will recruit heroin dependent persons from NYC jails who are soon-to-be-released, not accessing opioid agonist pharmacotherapy, with lowered tolerance due to incarceration, and extremely likely to relapse and risk accidental overdose at release. All N=40 participants receive a two-session, individual psychosocial intervention, Motivational Interviewing. Half (n=20) will be randomized to pre-release treatment with XR-NTX. Immediately and one month following release, participants will be offered continued psychosocial and medication-assisted treatment (naltrexone, buprenorphine, or methadone) at Bellevue Hospital, including a second XR-NTX dose among XR-NTX arm participants. The primary outcome is relapse to sustained opioid use during the first 30 days post-release. We hypothesize an XR-NTX arm will report significantly lower rates of sustained opioid relapse following release.

ELIGIBILITY:
Inclusion Criteria:

* Adults incarcerated in NYC jails with known release date
* DSM-IV criteria for current opioid dependence
* No current agonist (methadone, buprenorphine) treatment
* Currently opioid free by history ('detoxed') and with a negative urine for all opioids
* General good health as determined by complete medical interview and physical examination
* Age 18-60 years.

Exclusion Criteria:

* History of liver failure, cirrhosis, or recent liver function test levels greater than three times normal
* Pregnancy, lactation, or planning conception
* Active medical illness that might make participation hazardous
* Untreated psychiatric disorder
* History of allergic reaction to naltrexone, PLG (polylactide co-glycolide), carboxymethylcellulose, or any other components of the diluent.
* Current chronic pain condition treated with opioids.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Lee, MD MSc, Principal Investigator — NYU School of Medicine
Locations (2):
- United States (2):
  - New York University School of Medicine, New York, New York
  - New York City Department of Correction, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kornor H, Lobmaier PPK, Kunoe N. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2025 May 9;5(5):CD006140. doi: 10.1002/14651858.CD006140.pub3. PMID 40342086
- [Derived] Lee JD, McDonald R, Grossman E, McNeely J, Laska E, Rotrosen J, Gourevitch MN. Opioid treatment at release from jail using extended-release naltrexone: a pilot proof-of-concept randomized effectiveness trial. Addiction. 2015 Jun;110(6):1008-14. doi: 10.1111/add.12894. Epub 2015 Apr 5. PMID 25703440

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of participants took place at NYC jail medical clinics (Rikers Island; EMTC, RMSC) with follow-up visits taking place at Bellevue Hospital. The last participant completed in June 2013.
Pre-assignment Details: Of the 48 consented participants enrolled into study between January 2010-May 2013, 34 were randomized into one of two trial arms, with n=17 to Extended-Release Naltrexone arm and n=17 to the Motivational Enhancement Counseling Only arm (treatment-as-usual).
Period: Overall Study
Arm/Group | Extended-release Naltrexone (XR-NTX) | Motivational Enhancement Counseling Only
Started | 17 | 17
Completed | 12 | 11
Not Completed | 5 | 6
Not completed — Lost to Follow-up | 5 | 6

BASELINE CHARACTERISTICS:
Population: Baseline analysis determined based on: (1) successful randomization into one of two treatment arms (ETAU;XR-NTX) and (2) actual release from jail back to the community. One participant who successfully randomized to XR-NTX was never released from jail custody and was instead sent to prison and therefore excluded from final analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended-release Naltrexone (XR-NTX) | Motivational Enhancement Counseling Only | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 17 | 33
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 40 [26 to 52] | 47 [39 to 58] | 44 [26 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 17 | 33
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Post-Release Opioid Relapse
Description: Post-release opioid relapse at week 4, measured by self-report (Time Line Follow Back) and urine toxicologies, and defined as ≥10 of 28 days of self-reported opioid misuse following jail release or two or three positive of the three urine samples during weeks 2, 3 and 4. A single positive or missing urine result counted as 7 opioid misuse days.
Time Frame: Four weeks post-release
Population: One XR-NTX participant randomized was excluded from final data analysis due to the fact he was never released from jail to community, so primary outcome (post-release opioid relapse) could not be measured.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Extended-release Naltrexone (XR-NTX) | Motivational Enhancement Counseling Only
Number analyzed (Participants) | 16 | 17
participants | 6 [1 to 16] | 15 [1 to 17]

2. Secondary Outcome: Participation in Community Drug Treatment Post-release
Description: This secondary outcome tracks community drug treatment initiation four weeks post-release from jail. Measured by self-report community drug treatment initiation at week 4 study visit.
Time Frame: Four weeks post-release
Population: One XR-NTX participant who was randomized was excluded from final data analysis because he was never released from jail to community.
Measure: Number; unit: percentage of participants
Arm/Group | Extended-release Naltrexone (XR-NTX) | Motivational Enhancement Counseling Only
Number analyzed (Participants) | 16 | 17
percentage of participants | 19 | 12

3. Secondary Outcome: Any Opioid Use Post-release
Description: Counts of any opioid use, defined as self-reported ≥ 1 day of heroin or other opioid use as measured by the Timeline Follow-Back assessment during the first 4 weeks post-release.
Time Frame: Four weeks post-release
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Extended-release Naltrexone (XR-NTX) | Motivational Enhancement Counseling Only
Number analyzed (Participants) | 16 | 17
percentage of participants | 17 | 82

4. Secondary Outcome: Injection Drug Use Post-release
Description: This secondary outcome tracks any injection drug use and frequency of injection drug use in the four weeks following release from jail.
Time Frame: Four weeks post-release
Measure: Number; unit: percentage of participants by arm
Arm/Group | Extended-release Naltrexone (XR-NTX) | Motivational Enhancement Counseling Only
Number analyzed (Participants) | 16 | 17
percentage of participants by arm | 25 | 6

5. Secondary Outcome: Accidental Drug Overdose
Description: Accidental drug overdose is defined as patient self-report of any event consistent with over-sedation or respiratory suppression following ingestion of alcohol, prescription, or illicit drugs.
Time Frame: Four weeks post-release
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Extended-release Naltrexone (XR-NTX) | Motivational Enhancement Counseling Only
Number analyzed (Participants) | 16 | 17
participants | 0 | 0

6. Secondary Outcome: Adverse Events and Serious Adverse Events
Description: AEs and SAEs per standard definitions will be measured by self-report.
Time Frame: Eight weeks post-release
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Extended-release Naltrexone (XR-NTX) | Motivational Enhancement Counseling Only
Number analyzed (Participants) | 16 | 17
participants | 5 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events collected during 8 weeks post-release.
Arm/Group | Extended-release Naltrexone (XR-NTX) | Motivational Enhancement Counseling Only
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 5/16 | 1/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended-release Naltrexone (XR-NTX) (N=16) | Motivational Enhancement Counseling Only (N=17)
Anticipated XR-NTX Symptoms (General disorders) | 4 (4) | 0 (0) — Anticipated XR-NTX Symptoms including nausea, upset stomach, injection site soreness, dizziness, headache, and other flu-like symptoms.
Shoulder Seperation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Respiratory Problems (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations of this pilot study are: small sample size, no females enrolled in study, and no placebo control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No